CLINICAL TRIAL: NCT06362889
Title: An Exploratory Study to Evaluate the Safety and Efficacy of Microneedling With Cannabidiol (CBD) and Hempseed Oil for Treating Acne Vulgaris
Brief Title: Evaluating Microneedling With CBD and Hempseed Oil for Acne Vulgaris Safety and Efficacy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rejuva Medical Aesthetics (Other)
Collaborators: HealMD, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HealMD-CBD-1
Record Dates: First submitted 2024-04-05; First posted 2024-04-12 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Acne Vulgaris (Disorder)
MeSH Terms: conditions — Acne Vulgaris | interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Microneedling with CBD oil (Experimental): All subjects will receive microneedling with CBD oil.At the baseline visit, the subject will undergo treatment by the principal investigator or subinvestigator. 3 days from the treatment visit, a phone call visit will be placed to assess any safety events and adherence to protocol guidelines. Day 21 visit, several assessments will be recorded and if no adverse events are reported related to the study device and/or procedure, a second treatment will be performed. After 3 days from the treatment visit, a phone call will be placed to assess any safety events. Subjects will have subjective assessments and photographs taken at all visits. At day 42, the subject will return for a third treatment if no adverse events related to the study device and/or procedure are reported. After 3 days from the treatment visit, a phone call will be placed to assess any safety events. On day 63,no treatment to be performed, only a safety assessment, standardized assessments/questionnaires and photography.
  Interventions: Combination Product: Microneedling with CBD

INTERVENTIONS:
Combination Product: Microneedling with CBD — Cannabidiol (CBD) Isolate- 90-100mg / 1mL of carrier oil Organic Hemp Seed Oil- used as carrier oil for CBD isolate in Combination with Microneedling Device

SUMMARY:
This is a prospective, single center, open label study to assess the safety and effectiveness of microneedling with CBD and hempseed oil for the treatment of moderate to severe acne in adults 22-years of age or older.The objective of this exploratory study is to evaluate the safety and efficacy of HealMD's CBD with hempseed oil to reduce the appearance of moderate to severe facial acne.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female, 22 years of age or older. Females of childbearing potential must agree to the use of a reliable method of contraception throughout the study.
* Have a Global Acne Severity Scale Score of 3 (Moderate), 4 (Severe), or 5 (Very severe).
* Have no plans to begin a new skincare routine or medical treatment program (Accutane) through the course of the study.
* Willing to abstain from any aesthetic or surgical procedure in the treatment area for the duration of the study.

Exclusion Criteria:

* Significant history or current evidence of any uncontrolled chronic or serious disease or medical condition that would, in the judgment of the investigator, would put the subject at undue risk or compromise the study assessments.
* Employees of the Investigator or research center or their immediate family members.
* Inability to understand the requirements of the study and the relative information and are unable or not willing to comply with the study protocol.
* The use of Accutane (Isotretinoin) within 6-months.
* The use of topical or oral therapies that include benzoyl peroxide, azelaic acid, salicylic acid, and hydroquinone 30 days prior to study entry.
* Exposure to any other investigational drug/device within 30 days prior to study entry.
* Sunburned at time of anticipated treatment. Subject must also be willing to avoid significant sun exposure throughout participation
* Recent facial plastic surgery, aesthetic treatment, or dermatological treatment at treatment sites that would interfere with ability to receive microneedling.
* Facial hair that would interfere with the visualization of treatment sites.
* Subject with abnormal vision assessments.
* Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol (e.g. due to alcoholism, drug dependency, mental incapacity) in the opinion of the investigator.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoints | through study completion, approximately 70 days
  Reduction in the Global Acne Severity Scale (GAS) grade by Primary Investigator Reduction in the GAS grade by the Subject

SECONDARY OUTCOMES:
Secondary efficacy endpoints | through study completion, approximately 70 days
  Improvement in the appearance of acne vulgaris papules and comedones in standardized photographs Monitoring for Adverse Events and Serious Adverse Events at all study visits

CONTACTS AND LOCATIONS:
Overall Officials: Kian Karimi, MD, Principal Investigator — Rejuva Medical Aesthetics
Locations (1):
- Rejuva Medical Aesthetics, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The Data will be made available within 6 months of the study's conclusion, and will remain available for at least 5 years.
Access Criteria: Signing a data use agreement.

REFERENCES:
- [Background] Blaskovich MAT, Kavanagh AM, Elliott AG, Zhang B, Ramu S, Amado M, Lowe GJ, Hinton AO, Pham DMT, Zuegg J, Beare N, Quach D, Sharp MD, Pogliano J, Rogers AP, Lyras D, Tan L, West NP, Crawford DW, Peterson ML, Callahan M, Thurn M. The antimicrobial potential of cannabidiol. Commun Biol. 2021 Jan 19;4(1):7. doi: 10.1038/s42003-020-01530-y. PMID 33469147
- [Background] Peyravian N, Deo S, Daunert S, Jimenez JJ. The Anti-Inflammatory Effects of Cannabidiol (CBD) on Acne. J Inflamm Res. 2022 May 3;15:2795-2801. doi: 10.2147/JIR.S355489. eCollection 2022. PMID 35535052
- [Background] Atalay S, Jarocka-Karpowicz I, Skrzydlewska E. Antioxidative and Anti-Inflammatory Properties of Cannabidiol. Antioxidants (Basel). 2019 Dec 25;9(1):21. doi: 10.3390/antiox9010021. PMID 31881765
- [Background] Nachnani R, Raup-Konsavage WM, Vrana KE. The Pharmacological Case for Cannabigerol. J Pharmacol Exp Ther. 2021 Feb;376(2):204-212. doi: 10.1124/jpet.120.000340. Epub 2020 Nov 9. PMID 33168643
- [Background] Muller C, Morales P, Reggio PH. Cannabinoid Ligands Targeting TRP Channels. Front Mol Neurosci. 2019 Jan 15;11:487. doi: 10.3389/fnmol.2018.00487. eCollection 2018. PMID 30697147
- [Background] Huang T, Xu T, Wang Y, Zhou Y, Yu D, Wang Z, He L, Chen Z, Zhang Y, Davidson D, Dai Y, Hang C, Liu X, Yan C. Cannabidiol inhibits human glioma by induction of lethal mitophagy through activating TRPV4. Autophagy. 2021 Nov;17(11):3592-3606. doi: 10.1080/15548627.2021.1885203. Epub 2021 Feb 25. PMID 33629929
- [Background] Olah A, Toth BI, Borbiro I, Sugawara K, Szollosi AG, Czifra G, Pal B, Ambrus L, Kloepper J, Camera E, Ludovici M, Picardo M, Voets T, Zouboulis CC, Paus R, Biro T. Cannabidiol exerts sebostatic and antiinflammatory effects on human sebocytes. J Clin Invest. 2014 Sep;124(9):3713-24. doi: 10.1172/JCI64628. Epub 2014 Jul 25. PMID 25061872
- [Background] Alqam ML, Jones BC, Hitchcock TM. Study to determine the safety and efficacy of microneedling as an effective treatment for acne vulgaris. Skin Health Dis. 2023 Jul 5;3(5):e264. doi: 10.1002/ski2.264. eCollection 2023 Oct. PMID 37799356
- [Background] Land MH, Toth ML, MacNair L, Vanapalli SA, Lefever TW, Peters EN, Bonn-Miller MO. Effect of Cannabidiol on the Long-Term Toxicity and Lifespan in the Preclinical Model Caenorhabditis elegans. Cannabis Cannabinoid Res. 2021 Dec;6(6):522-527. doi: 10.1089/can.2020.0103. Epub 2020 Nov 20. PMID 33998871
- [Background] Cerne K. Toxicological properties of Delta9-tetrahydrocannabinol and cannabidiol. Arh Hig Rada Toksikol. 2020 Mar 1;71(1):1-11. doi: 10.2478/aiht-2020-71-3301. PMID 32597140